CLINICAL TRIAL: NCT06000137
Title: The Comparison of the Analgesic Effects of Dezocine and Sufentanil in Patient-controlled Analgesia After Laryngectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: dezocine and sufentanil
Record Dates: First submitted 2023-05-04; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Patient-controlled Analgesia
Keywords: dezocine; sufentanil; laryngectomy; patient-controlled analgesia
MeSH Terms: interventions — dezocine; Sufentanil; Flurbiprofen; Granisetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group S (Experimental): sufentanil 2μg/kg + flurbiprofen 250mg+granisetron 6mg
  Interventions: Drug: Sufentanil injection; Drug: Flurbiprofen; Drug: Granisetron Injection
- group D1 (Active Comparator): dezocine 0.5mg/kg + flurbiprofen 250mg+granisetron 6mg
  Interventions: Drug: Dezocine; Drug: Flurbiprofen; Drug: Granisetron Injection
- group D2 (Active Comparator): dezocine 0.6mg/kg + flurbiprofen 250mg+granisetron 6mg
  Interventions: Drug: Dezocine; Drug: Flurbiprofen; Drug: Granisetron Injection

INTERVENTIONS:
Drug: Dezocine — dezocine for patient-controlled analgesia
  Arms: group D1; group D2
Drug: Sufentanil injection — sufentanil for patient-controlled analgesia
  Other Names: sufentanil
  Arms: group S
Drug: Flurbiprofen — Flurbiprofen for patient-controlled analgesia
Drug: Granisetron Injection — granisetron has antiemetic function.
  Other Names: granisetron

SUMMARY:
Laryngeal cancer is one of the most common tumors in otolaryngology. In China, it accounts for 1-5% of all malignancies and has an incidence of 1.13 per 100,000. Surgical resection is the most important treatment for patients who are not candidates for chemoradiotherapy or refuse chemoradiotherapy. The types of surgery include total and partial laryngectomy. Patients with laryngeal cancer often face multiple physical and psychiatric changes after surgery, such as daily large sputum production accompanied by cough, cleaning care of the air incision, fatigue, and sleep disturbances. Some patients do not actively exclude secretions due to pain, and the formation of sputum plugs causes lung inflammation, which is not conducive to postoperative recovery. Good postoperative pain management is beneficial to shorten the length of hospital stay and reduce mortality. Sufentanil is most commonly used for postoperative analgesia and has good analgesic effect, but there are some adverse effects, such as dizziness, nausea and vomiting, urinary retention, skin itching, respiratory depression, etc. As a new type of analgesic, dezocine has been widely used in clinical practice with few adverse reactions to the respiratory and circulatory system, and its application to postoperative analgesia can significantly improve the immune activity. At present, there are not many studies on continuous analgesia of dezocine, mostly single-dose analgesia studies, this study for different doses of dezocine for the postoperative analgesic effect of laryngeal cancer patients, compared with the current classic opioid analgesics, to provide a new scheme for clinical medication.

DETAILED DESCRIPTION:
Laryngeal cancer is one of the most common tumors in otolaryngology. In China, it accounts for 1-5% of all malignancies and has an incidence of 1.13 per 100,000. Surgical resection is the most important treatment for patients who are not candidates for chemoradiotherapy or refuse chemoradiotherapy. The types of surgery include total and partial laryngectomy. Patients with laryngeal cancer often face multiple physical and psychiatric changes after surgery, such as daily large sputum production accompanied by cough, cleaning care of the air incision, fatigue, and sleep disturbances. In patients with laryngeal cancer, large amounts of secretions can cause frequent coughing, even wheezing, and coughing can exacerbate the degree of postoperative pain. Some patients do not actively exclude secretions due to pain, and the formation of sputum plugs causes lung inflammation, which is not conducive to postoperative recovery. In addition, the inability to verbalize after laryngeal cancer surgery puts patients in a state of anxiety, which increases the degree of postoperative pain. Good postoperative pain management is beneficial to shorten the length of hospital stay and reduce mortality. Sufentanil is most commonly used for postoperative analgesia and has good analgesic effect, but there are some adverse effects, such as dizziness, nausea and vomiting, urinary retention, skin itching, respiratory depression, etc. As a new type of analgesic, dezocine has been widely used in clinical practice with few adverse reactions to the respiratory and circulatory system, and its application to postoperative analgesia can significantly improve the immune activity. At present, there are not many studies on continuous analgesia of dezocine, mostly single-dose analgesia studies, this study for different doses of dezocine for the postoperative analgesic effect of laryngeal cancer patients, compared with the current classic opioid analgesics, to provide a new scheme for clinical medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent elective partial laryngectomy
* American society of Anesthesiologists (ASA) physical status classification :Ⅰ~Ⅱ

Exclusion Criteria:

* chronic pain
* long-term use of analgesics
* allergy to perioperative medications
* previous postoperative nausea and vomiting

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-01-14 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
total | from the end of the surgery to 48 hours after surgery
  no pain =0, mild pain =1-3, moderate pain =4-6, and severe pain =7-10

SECONDARY OUTCOMES:
24 hours amount of drug | From the time of use postoperative analgesic to the time of 24 hours after the surgery
  the volume of postoperative analgesic in 24 hours after the surgery
48 hours pressing times of Patient-controlled Analgesia | From the time of use postoperative analgesic to the time of 48 hours after the surgery
  the times of press analgesia pump in 24 hours after the surgery
Visual Analogue Scale | at the time of 6 hours after the surgery
  no pain =0, mild pain =1-3, moderate pain =4-6, and severe pain =7-10
Visual Analogue Scale | at the time of 12 hours after the surgery
  no pain =0, mild pain =1-3, moderate pain =4-6, and severe pain =7-10
Visual Analogue Scale | at the time of 24 hours after the surgery
  no pain =0, mild pain =1-3, moderate pain =4-6, and severe pain =7-10
Visual Analogue Scale | at the time of 48 hours after the surgery
  no pain =0, mild pain =1-3, moderate pain =4-6, and severe pain =7-10
the incidence of nausea | from the time when patients use postoperative analgesic to the time when patients stop to use postoperative analgesic, assessed up to 48 hours
  the incidence of nausea
the incidence of vomiting | from the time when patients use postoperative analgesic to the time when patients stop to use postoperative analgesic, assessed up to 48 hours
  the incidence of vomiting
the incidence of dizziness | from the time when patients use postoperative analgesic to the time when patients stop to use postoperative analgesic, assessed up to 48 hours
  the incidence of dizziness
the incidence of urinary | from the time when patients use postoperative analgesic to the time when patients stop to use postoperative analgesic, assessed up to 48 hours
  the incidence of urinary
the incidence of respiratory depression | from the time when patients use postoperative analgesic to the time when patients stop to use postoperative analgesic, assessed up to 48 hours
  the incidence of respiratory depression

CONTACTS AND LOCATIONS:
Overall Officials: Jie Li, Study Chair — Fudan University
Locations (1):
- Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Budliger H, Prader A, Morscher E, Fendel H. [Round table discussion on bone age]. Radiologe. 1971 Aug;11(8):296-9. No abstract available. German. PMID 4329172
- [Background] Perry F, Parker RK, White PF, Clifford PA. Role of psychological factors in postoperative pain control and recovery with patient-controlled analgesia. Clin J Pain. 1994 Mar;10(1):57-63; discussion 82-5. doi: 10.1097/00002508-199403000-00008. PMID 8193445
- [Background] O'Brien JJ, Benfield P. Dezocine. A preliminary review of its pharmacodynamic and pharmacokinetic properties, and therapeutic efficacy. Drugs. 1989 Aug;38(2):226-48. doi: 10.2165/00003495-198938020-00005. PMID 2670517
- [Background] Wang YX, Mao XF, Li TF, Gong N, Zhang MZ. Dezocine exhibits antihypersensitivity activities in neuropathy through spinal mu-opioid receptor activation and norepinephrine reuptake inhibition. Sci Rep. 2017 Feb 23;7:43137. doi: 10.1038/srep43137. PMID 28230181
- [Background] Gharagozlou P, Demirci H, Clark JD, Lameh J. Activation profiles of opioid ligands in HEK cells expressing delta opioid receptors. BMC Neurosci. 2002 Nov 18;3:19. doi: 10.1186/1471-2202-3-19. Epub 2002 Nov 18. PMID 12437765
- [Background] Liu R, Huang XP, Yeliseev A, Xi J, Roth BL. Novel molecular targets of dezocine and their clinical implications. Anesthesiology. 2014 Mar;120(3):714-23. doi: 10.1097/ALN.0000000000000076. PMID 24263237
- [Background] Bian X, Zhou R, Yang Y, Li P, Hang Y, Hu Y, Yang L, Wen D. Divergent Effect of Dezocine, Morphine and Sufentanil on Intestinal Motor Function in Rats. Int J Med Sci. 2015 Oct 15;12(11):848-52. doi: 10.7150/ijms.12616. eCollection 2015. PMID 26640403
- [Background] Zhou X, Zhang C, Wang M, Yu L, Yan M. Dezocine for Preventing Postoperative Pain: A Meta-Analysis of Randomized Controlled Trials. PLoS One. 2015 Aug 19;10(8):e0136091. doi: 10.1371/journal.pone.0136091. eCollection 2015. PMID 26287536
- [Background] Wang C, Li L, Shen B, Jiang H, Yuan L, Shi D, Zhu J, Guo X, Li H. A multicenter randomized double-blind prospective study of the postoperative patient controlled intravenous analgesia effects of dezocine in elderly patients. Int J Clin Exp Med. 2014 Mar 15;7(3):530-9. eCollection 2014. PMID 24753745
- [Background] Zhou L, Zhang Y, Sun H, Hu R, Wang J, Xu G. Effect of preemptive dezocine before general anesthesia on postoperative analgesia in patients undergoing laparoscopic cholecystectomy: A prospective observational study. Medicine (Baltimore). 2018 Sep;97(39):e12533. doi: 10.1097/MD.0000000000012533. PMID 30278544